CLINICAL TRIAL: NCT02091362
Title: The Effect of LY2409021 on Blood Pressure and Pulse Rate, as Assessed by Ambulatory Blood Pressure Monitoring, in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study of LY2409021 on Blood Pressure and Pulse Rate in Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 15261; I1R-MC-GLDI (Other: Eli Lilly and Company); 2013-003834-33 (EudraCT Number)
Record Dates: First submitted 2014-03-18; First posted 2014-03-19 (Estimated); Results first posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — adomeglivant; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Single daily dose of placebo matching LY2409021 administered orally in 1 of 2 treatment periods.
  Interventions: Drug: Placebo; Drug: Metformin
- LY2409021 (Experimental): Single daily dose of 20 milligrams (mg) LY2409021 administered orally in 1 of 2 treatment periods.
  Interventions: Drug: LY2409021; Drug: Metformin

INTERVENTIONS:
Drug: LY2409021 — Administered orally
  Arms: LY2409021
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: Metformin — Administered as background therapy.

SUMMARY:
The main purpose of the trial is to determine the effect of a study drug known as LY2409021 on blood pressure and pulse rate in participants with type 2 diabetes mellitus (T2DM) when compared to placebo. The study has two periods. Each participant will receive LY2409021 or placebo in each period. At least 4 weeks will pass between periods. The study will last about 23 weeks for each participant. Participants may remain on stable dose metformin, as prescribed by their personal physician.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes mellitus (according to the World Health Organization diagnostic criteria) and use diet and exercise alone or in combination with a stable dose of metformin ( >/=1000 mg/day [or <1000 mg, if documented intolerance to 1000 mg or higher dosages] immediate-release metformin or extended-release metformin for at least 2 months before screening).
* Have glycated hemoglobin (HbA1c) values >/=6.5% and </=8.5%, as determined by the central laboratory at screening.
* Have mean blood pressures >90/60 millimeters of mercury (mm Hg) and <140/90 mm Hg at screening.
* If being treated for hypertension, are taking 3 or fewer antihypertensive medications and have been taking stable doses of the same medications for at least 1 month before screening.
* Stable body weights (±5%) for >/=3 months before screening.
* Body mass indexes >/=20 kilograms/meters squared (kg/m²) and <40 kg/m².
* In the investigator's opinion, are well motivated, capable, and willing to:

  * Reliably administer the oral study drug once daily;
  * Maintain a study diary;
  * Perform self-monitored blood glucose testing; and
  * Wear an ambulatory blood pressure monitoring device for at least 24 hours (on multiple occasions).
* Are women not of child-bearing potential due to:

  * Surgical sterilization, hysterectomy, or bilateral oophorectomy (at least 6 weeks postsurgery) or tubal ligation (confirmed by medical history); or
  * Menopause. Women with an intact uterus are deemed menopausal if they have a cessation of menses for at least 1 year with follicle stimulating hormone >40 milli-international units per milliliter (mIU/mL), are not taking hormones or oral contraceptives within 1 year, and are otherwise healthy.
* Males who are sexually active and/or have partners of child-bearing age must use reliable methods of birth control during the study and until 3 months after the last doses of study medication. These requirements do not apply if a participant or his partner has been surgically sterilized or is not between menarche and 1 year postmenopausal.

Exclusion Criteria:

* Have severe gastrointestinal disease that may significantly affect gastric emptying or motility.
* Previous histories or active diagnoses of pancreatitis.
* Acute or chronic hepatitis, signs or symptoms of any other liver disease, or alanine aminotransferase (ALT) level greater than 2.5 times the upper limit of normal (ULN).
* Elevated total bilirubin (greater than 2 times ULN), clinically suspicious signs or symptoms of cirrhosis or history of cirrhosis.
* Mean resting pulse rate (PR) less than 60 beats per minute (bpm) or greater than 100 bpm.
* Current diagnosis or personal history of neuroendocrine tumors, family history of any type of multiple endocrine neoplasia, or Von Hippel-Lindau disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (29):
- United States (15):
  - Advanced Clinical Research Institute, Anaheim, California
  - National Research Institute, Los Angeles, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Orange County Research Center, Tustin, California
  - University Clinical Investigators, Inc., Tustin, California
  - Berma Research, Fort Lauderdale, Florida
  - East Coast Clinical Research, Jacksonville, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - L-Marc Research Center, Louisville, Kentucky
  - Maine Research Associates, Auburn, Maine
  - Alzohaili Medical Consultants, Dearborn, Michigan
  - Premier Research, Trenton, New Jersey
  - Manhattan Medical Research, New York, New York
- Czechia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Holešov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krnov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pardubice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coatzacoalcos
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- Poland (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
- Puerto Rico (2):
  - Manati Center for Clinical Research Inc, Manatí
  - Consultorio Medico, San Juan

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2409021/Placebo: Period 1: Single daily dose of 20 milligrams (mg) LY2409021 administered orally for 6 weeks; Wash-out: 4 weeks; Period 2: Single daily dose of placebo administered orally for 6 weeks.
- Placebo/LY2409021: Period 1: Single daily dose of placebo administered orally for 6 weeks; Wash-out: 4 weeks; Period 2: Single daily dose of 20 milligrams (mg) LY2409021 administered orally for 6 weeks.
Period: Period 1
Arm/Group | LY2409021/Placebo | Placebo/LY2409021
Started | 133 | 137
Completed | 128 | 133
Not Completed | 5 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 2 | 0
Period: Wash-out
Arm/Group | LY2409021/Placebo | Placebo/LY2409021
Started | 128 | 133
Completed | 127 | 130
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2
Period: Period 2
Arm/Group | LY2409021/Placebo | Placebo/LY2409021
Started | 127 | 130
Completed | 125 | 128
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- LY2409021 20 mg: Period 1: Single daily dose of 20 mg LY2409021 administered orally for 6 Weeks; Wash-out: 4 weeks; Period 2: Single daily dose of placebo administered orally for 6 weeks.
- Placebo: Period 1: Single daily dose of placebo administered orally for 6 weeks; Wash-out: 4 weeks; Period 2: Single daily dose of 20 mg Ly2409021 administered orally for 6 weeks.
- Total: Total of all reporting groups
Arm/Group | LY2409021 20 mg | Placebo | Total
Number analyzed (Participants) | 133 | 137 | 270
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (8.9) | 57.2 (8.9) | 57.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 60 | 117
  Male | 76 | 77 | 153
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 63 | 62 | 125
  Not Hispanic or Latino | 61 | 69 | 130
  Unknown or Not Reported | 9 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 20 | 22 | 42
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 23 | 35
  White | 92 | 87 | 179
  More than one race | 7 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Czechia | 19 | 22 | 41
  United States | 72 | 74 | 146
  Poland | 18 | 18 | 36
  Mexico | 24 | 23 | 47
Diagnosis of Hypertension [Count of Participants; unit: Participants]
  Yes | 89 | 93 | 182
  No | 44 | 44 | 88
Hemoglobin A1c (HBA1c) [Count of Participants; unit: Participants]
  ≥ 7.5 % | 49 | 51 | 100
  < 7.5% | 84 | 86 | 170

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 6 Weeks in Mean 24-Hour Systolic Blood Pressure
Description: Systolic blood pressure obtained from Ambulatory Blood Pressure Monitoring (ABPM).
Time Frame: Baseline, 6 Weeks
Population: Modified intent-to-treat (mITT) population consisting of all randomized subjects who received at least one dose of study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Groups:
- LY2409021 20 mg: Single daily dose of 20 milligrams (mg) LY2409021 administered orally in 1 of 2 treatment periods
Arm/Group | LY2409021 20 mg | Placebo
Number analyzed (Participants) | 241 | 239
mmHg | 2.79 [1.62 to 3.95] | 0.53 [-0.70 to 1.76]
Statistical Analysis 1: Comparison: LY2409021 20 mg vs Placebo; Test type: Superiority or Other; p < .001, Mixed Models Analysis; LS Mean Difference = 2.26, 95% CI 2-sided [1.11 to 3.40]

2. Secondary Outcome: Change From Baseline to 6 Weeks in Mean 24-Hour Diastolic Blood Pressure
Description: Diastolic blood pressure obtained from Ambulatory Blood Pressure Monitoring (ABPM). LS Mean of treatment differences, adjusted for country, diagnosis of hypertension, sequence, treatment, period, time within period, treatment by time within period interaction, and the baseline measurement as covariate.
Time Frame: Baseline, 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | LY2409021 20 mg | Placebo
Number analyzed (Participants) | 241 | 239
mmHg | 1.37 [0.61 to 2.14] | 0.00 [-0.76 to 0.77]
Statistical Analysis 1: Comparison: LY2409021 20 mg vs Placebo; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; LS Mean Difference = 1.37, 95% CI 2-sided [0.66 to 2.08]

3. Secondary Outcome: Change From Baseline to 6 Weeks in Mean 24-Hour, Daytime, and Nighttime Peripheral Pulse Rate
Description: Pulse rate obtained from Ambulatory Blood Pressure Monitoring (ABPM). LS Mean of treatment differences, adjusted for country, diagnosis of hypertension, sequence, treatment, period, time within period, treatment by time within period interaction, and the baseline measurement as covariate.
Time Frame: Baseline, 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: beats/minute
Arm/Group | LY2409021 20 mg | Placebo
Number analyzed (Participants) | 241 | 239
beats/minute
  24 Hour Pulse Rate | 0.46 [-0.46 to 1.37] | 0.43 [-0.53 to 1.40]
  Mean Daytime Pulse Rate | 0.74 [-0.26 to 1.75] | 0.56 [-0.48 to 1.61]
  Mean Nighttime Pulse Rate | -0.39 [-1.35 to 0.57] | -0.04 [-1.03 to 0.96]

4. Secondary Outcome: Change From Baseline to 6 Weeks in Mean 24-Hour, Daytime, and Nighttime Pulse Pressures
Description: Pulse Pressures obtained from Ambulatory Blood Pressure Monitoring (ABPM). LS Mean of treatment differences, adjusted for country, diagnosis of hypertension, sequence, treatment, period, time within period, treatment by time within period interaction, and the baseline measurement as covariate.
Time Frame: Baseline, 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | LY2409021 20 mg | Placebo
Number analyzed (Participants) | 241 | 239
mmHg
  24-Hour Pulse Pressure | 1.51 [0.76 to 2.25] | 0.62 [-0.13 to 1.38]
  Daytime Pulse Pressure | 1.49 [0.68 to 2.29] | 0.54 [-0.29 to 1.38]
  Nighttime Pulse Pressure | 1.51 [0.69 to 2.32] | 0.80 [0.00 to 1.60]

5. Secondary Outcome: Change From Baseline to 6 Weeks in Mean 24-Hour, Daytime, and Nighttime Mean Arterial Pressures (MAP)
Description: Mean Arterial Pressures obtained from Ambulatory Blood Pressure Monitoring (ABPM). LS Mean of treatment differences, adjusted for country, diagnosis of hypertension, sequence, treatment, period, time within period, treatment by time within period interaction, and the baseline measurement as covariate.
Time Frame: Baseline, 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | LY2409021 20 mg | Placebo
Number analyzed (Participants) | 241 | 239
mmHg
  24 Hour MAP | 1.83 [0.99 to 2.68] | 0.17 [-0.71 to 1.04]
  Daytime MAP | 2.04 [1.14 to 2.94] | 0.08 [-0.86 to 1.03]
  Nighttime MAP | 1.31 [0.33 to 2.29] | 0.33 [-0.68 to 1.33]

6. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: LS Mean of treatment differences, adjusted for country, diagnosis of hypertension, sequence, treatment, period, time within period, treatment by time within period interaction, and the baseline measurement as covariate.
Time Frame: Baseline, 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of HbA1c
Arm/Group | LY2409021 20 mg | Placebo
Number analyzed (Participants) | 241 | 239
percentage of HbA1c | -0.65 [-0.72 to -0.58] | -0.16 [-0.23 to -0.08]

7. Secondary Outcome: Population Pharmacokinetics: Apparent Clearance of LY2409021
Description: Population pharmacokinetic parameter apparent clearance (CL/F) is the apparent volume of the body fluid cleared of the drug per unit of time and was estimated by modeling of LY2409021 plasma concentration data from all LY2409021 groups.
Time Frame: Days 7, 21, 42, 70, 77, 91, 112, 140; 15 minute Predose and Days 7 and 77: 1 hour Postdose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/hr)
Arm/Group | LY2409021 20 mg
Number analyzed (Participants) | 249
Liter per hour (L/hr) | 0.406 (30.7)

8. Secondary Outcome: Population Pharmacokinetics: Apparent Volume of Distribution of LY2409021
Description: Population pharmacokinetic parameter, apparent volume of distribution (V/F) is a theoretical volume that a drug would have to occupy (if it were uniformly distributed), to provide the same concentration as it currently is in blood plasma. Apparent volume of distribution (V/F) was estimated by modeling of LY2409021 plasma concentration data from all LY2409021 groups.
Time Frame: Days 7, 21, 42, 70, 77, 91, 112, 140; Predose and Days 7 and 77: 1 hour Postdose.
Population: All randomized participants who received at least 1 one dose of study drug and had at least one measureable drug concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | LY2409021 20 mg
Number analyzed (Participants) | 249
Liters | 36.7 (23.2)

ADVERSE EVENTS:
Groups:
- LY2409021 20 mg: AEs (Adverse Event) from Period 1 and 2 combined from LY2409021 20 mg administration
- Placebo: AEs from Period 1 and 2 combined from placebo administration.
- Wash-out: All AEs included during wash-out period.
- Follow-up: All AEs from follow-up period.
Arm/Group | LY2409021 20 mg | Placebo | Wash-out | Follow-up
Serious Adverse Events (participants affected / at risk) | 4/258 | 2/256 | 2/249 | 4/253
Other Adverse Events (participants affected / at risk) | 49/258 | 32/256 | 25/249 | 30/253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2409021 20 mg (N=258) | Placebo (N=256) | Wash-out (N=249) | Follow-up (N=253)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2409021 20 mg (N=258) | Placebo (N=256) | Wash-out (N=249) | Follow-up (N=253)
Abdominal discomfort (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 3 (3) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 3 (3) | 3 (3)
Alanine aminotransferase increased (Investigations) | 12 (12) | 1 (1) | 4 (4) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 2 (2) | 2 (2) | 3 (3)
Blood pressure diastolic increased (Investigations) | 3 (3) | 3 (3) | 2 (2) | 2 (2)
Heart rate decreased (Investigations) | 3 (4) | 2 (3) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 4 (6) | 3 (3) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) | 3 (5) | 3 (3)
Dizziness (Nervous system disorders) | 3 (4) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 4 (5) | 4 (4) | 2 (3) | 3 (5)
Hypertension (Vascular disorders) | 2 (2) | 3 (3) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days